CLINICAL TRIAL: NCT01543425
Title: Status of the Hypothalamic-pituitary-gonado- Adrenal Axis (HHSG) in Patients With Neuropathic Pain
Brief Title: Adrenocorticotropic Axis and Neuropathic Pain
Acronym: HORMONES
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: CHU-0116
Record Dates: First submitted 2012-02-28; First posted 2012-03-05 (Estimated); Last update posted 2013-05-14 (Estimated); Status verified 2013-05

CONDITIONS: Neuropathic Pain
Keywords: Neuropathic Pain; Adenocorticotrophic axis; Psychological state
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — Day of inclusion: Blood sample for analysis of several hormones (cortisol, ACTH, SHBG, total testostérone et S-DHEA, βœstradiol et progestérone for women, LH, FSH).
  Day +1: salivary samples (at wake-up, 30 minutes after wake-up, at lunch, at 06:00 pm and before sleep).
  Day +2: salivary samples (at wake-up, 30 minutes after wake-up).

SUMMARY:
Chronic pain is often associated with a chronic stress and HHSG axis plays a pivotal role in maintaining homeostasis. The literature reports that pain in patients treated with opioids, significant changes are taking place in this axis with a collapse in hormone concentrations that are correlated with the decline on tests of quality of life and psychological testing. The investigators hypothesis is that this "endocrinopathy" could also be present in patients treated for neuropathic pain with other drug classes as opiates (antidepressants, antiepileptics), and may explain, at least in part, the impairement of the quality of life of these patients.

DETAILED DESCRIPTION:
Day of inclusion: Blood sample for analysis of several hormones (cortisol, ACTH, SHBG, total testostérone et S-DHEA, βœstradiol et progestérone for women, LH, FSH).

Day +1: salivary samples (at wake-up, 30 minutes after wake-up, at lunch, at 06:00 pm and before sleep).

Day +2: salivary samples (at wake-up, 30 minutes after wake-up).

ELIGIBILITY:
Inclusion Criteria:

* Group of patients
* Patients older than 18 years,
* Male or Female with BMI between 18 and 35,
* Patients with chronic neuropathic pain for more than six months, except to diabetes or central neuropathic pain
* Patients receiving systemic therapy for treating chronic neuropathic pain such as antidepressants, anticonvulsants or opiates for at least 6 months.

Group of healthy volunteers

* non-painful healthy volunteers matched by age, sex, BMI and menopausal status for women,
* Free of analgesics within 8 days before the test,
* Aged over 18 years,
* Male or Female,

Exclusion Criteria:

* Subjects with a medical history and / or surgical judged by the investigator or his representative as being incompatible with the test
* Patients treated only by topical treatment (lidocaine patch only for example)
* Pateints receiving corticosteroid treatment at the time of enrollment, or who received such treatment during the last 6 months (regardless of the dosage form and dosage),
* Inflammatory and evolutive pathology requiring long term treatment,
* Type 2 diabetes,
* Postmenopausal women with replacement therapy,
* Weight change of more than 5% within 3 months before the study,
* BMI <18 or> 35,

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients older than 18 years,
  * Male or Female with BMI between 18 and 35,
  * Patients with chronic neuropathic pain for more than six months, except to diabetes or central neuropathic pain
  * Patients receiving systemic therapy for treating chronic neuropathic pain such as antidepressants, anticonvulsants or opiates for at least 6 months.
  Group of healthy volunteers
  * non-painful healthy volunteers matched by age, sex, BMI and menopausal status for women,
  * Free of analgesics within 8 days before the test,
  * Aged over 18 years,
  * Male or Female,
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2012-03; Primary Completion 2013-02 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
hormonal status of neuropathic patients (blood sample ) | at day 0

SECONDARY OUTCOMES:
hormonal status of neuropathic patients, salivary sample | at day 1 and 2
Collection of different drug classes (antidepressants, antiepileptics, opioids) | at day 0,
scale anxiety / depression HAD | at day 0
cognitive state | at day 0,
SF36 questionnaire | at day 0
physical activity questionnaire (IPAQ) | at day 0
body mass index (BMI / Impedancemetry) | at day 0
waist circumference | at day 0

CONTACTS AND LOCATIONS:
Overall Officials: Gisèle PICKERING, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Corriger A, Duclos M, Corcuff JB, Lambert C, Marceau G, Sapin V, Macian N, Roux D, Pereira B, Pickering G. Hormonal Status and Cognitivo-Emotional Profile in Real-Life Patients With Neuropathic Pain: A Case Control Study. Pain Pract. 2019 Sep;19(7):703-714. doi: 10.1111/papr.12800. Epub 2019 Jun 27. PMID 31127700